CLINICAL TRIAL: NCT04142177
Title: CSP #2009 - Sequential and Comparative Evaluation of Pain Treatment Effectiveness Response: The SCEPTER Trial
Brief Title: Sequential and Comparative Evaluation of Pain Treatment Effectiveness Response
Acronym: SCEPTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2009
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; severe low back pain; pain; non-pharmacological treatment; self-management; physical therapy; exercise; yoga; cognitive behavioral therapy; spinal manipulation therapy
MeSH Terms: conditions — Low Back Pain; Pain; Motor Activity | interventions — pain ease refrigerant; Cognitive Behavioral Therapy; Yoga

STUDY DESIGN:
Intervention Model Description: sequential randomized, pragmatic, 2-step comparative effectiveness study design
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded study. The participants, Local Site Investigators (LSIs) and Site Coordinators will have the information on participant treatment assignment. Centralized Outcome Assessors (COAs) who collect primary and secondary outcome measures over the phone will be blinded to treatment assignment. The study team who manage the day-to-day study operations (including Study Chairs, National Study Coordinator, and study team members at Cooperative Studies Program Coordinating Centers [CSPCC] and Clinical Research Pharmacy Coordinating Centers [CRPCC] may have information on specific individual participant treatment assignment only when the information is needed to perform their work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Internet-based pain self-management program (Active Comparator): Internet-based treatment (Step 1 Treatment)
  Interventions: Other: Pain EASE
- Enhanced Physical Therapy (Active Comparator): Intervention that combines the internet-based pain self-management program with tailored exercise and physical activity guided by a physical therapist (Step 1 treatment)
  Interventions: Other: Pain EASE; Procedure: Tailored exercise
- Continued Care and Active Monitoring (CCAM) (Placebo Comparator): CCAM will not be standardized keeping in line with the pragmatic nature of this trial. CCAM may be variable across sites and for individual participants reflecting de facto clinical practice for cLBP. Clinical practice may involve pharmacological and non-pharmacological treatments for cLBP. Current analgesics (including opioids, acetaminophen, NSAIDs, topical analgesics (capsaicin), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, skeletal muscle relaxants, and alpha-2-delta ligands (gabapentin-like drugs)) and non-pharmacological treatments may be continued by participants. CCAM participants will be encouraged to discuss pain problems with their treating physician, but not begin new treatments if possible. Patients will specifically be discouraged from starting CBT, chiropractic, or yoga. Other than this, there will be no attempt by study personnel to influence pain management (Step 1 Treatment)
  Interventions: Other: Continued Care and Active Monitoring
- Cognitive Behavioral Therapy (CBT) (Active Comparator): Participants randomized to CBT in Step 2 will receive treatment with a trained therapist using the VA's CBT-chronic pain (CBT-CP) protocol involving one planning session and 9 treatment sessions (10 total) over 3 months (Step 2 Treatment).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Spinal Manipulation Therapy (SMT) (Active Comparator): After examination by a qualified Doctor of Chiropractic (DC), a SMT intervention consisting of up to 10 sessions over 3 months will be designed focusing on spinal manipulation and/or mobilization of the lower thoracic, lumbar and/or sacroiliac joints. Adjunctive use of myofascial and/or stretching techniques are allowed as they are commonly used along with SMT, and can be considered a standard accompaniment to SMT (Step 2 Treatment).
  Interventions: Procedure: Spinal Manipulation Therapy (SMT)
- Yoga (Active Comparator): The Yoga for Veterans with cLBP program consists of up to 10 weekly, 60-minute instructor-led sessions along with 15-20 minutes of yoga practiced at home each non-session day. The initial session is 75 minutes (15 minutes longer than the other sessions). The yoga program can be considered classical hatha yoga with influences from Iyengar and Viniyoga yoga. These styles emphasize modifications and adaptations including the use of props such as straps and blocks to minimize the risk of injury and make the poses accessible to people with health problems and limitations (Iyengar, 1979). The instructor leads participants through a series of 23 yoga poses (32 total variations) at a slow-moderate pace (Step 2 Treatment).
  Interventions: Procedure: Yoga

INTERVENTIONS:
Other: Pain EASE — The internet-based pain self-management program consists of open access to the Pain EASE program (Pain E-health for Activity, Skills, and Education) for the duration of participation in the trial. Pain EASE has 10 pain coping skill modules: pain education, setting personal goals, planning meaningful activities, physical activity (stretching, body mechanics, and a pedometer-based walking program), relaxation, developing healthy thinking patterns, pacing and problem-solving, improving sleep, effective communication, and future planning.
  Arms: Enhanced Physical Therapy; Internet-based pain self-management program
Procedure: Tailored exercise — Findings from the initial examination and the Keele STarT Back Screening Tool (Hill, et al., 2011) will be used by the physical therapist to guide and tailor the intervention to individual participants which will involve up to 8 treatment sessions with ongoing home exercise. For most participants, exercise and physical activity will focus on walking in addition to motor control and stabilization exercises for the low back with flexibility exercises when lumbar spine stiffness is present.
  Arms: Enhanced Physical Therapy
Other: Continued Care and Active Monitoring — CCAM will not be standardized keeping in line with the pragmatic nature of this trial. CCAM may be variable across sites and for individual participants reflecting de facto clinical practice for cLBP. Clinical practice may involve pharmacological and non-pharmacological treatments for cLBP. Current analgesics (including opioids, acetaminophen, NSAIDs, topical analgesics (capsaicin), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, skeletal muscle relaxants, and alpha-2-delta ligands (gabapentin-like drugs)) and non-pharmacological treatments may be continued by participants. CCAM participants will be encouraged to discuss pain problems with their treating physician, but not begin new treatments if possible. Patients will specifically be discouraged from starting CBT, chiropractic, or yoga. Other than this, there will be no attempt by study personnel to influence pain management.
  Arms: Continued Care and Active Monitoring (CCAM)
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants randomized to CBT in Step 2 will receive treatment with a trained therapist using the VA's CBT-chronic pain (CBT-CP) protocol involving one planning session and 9 treatment sessions (10 total) over 3 months. The VA's CBT-CP protocol consists of 11 core CBT-CP modules that can be completed in up to 10 sessions. Weekly, individual sessions of 45-50 minutes are recommended, although it is recognized that bi-weekly or other arrangements are often made to fit practical needs.
  Arms: Cognitive Behavioral Therapy (CBT)
Procedure: Spinal Manipulation Therapy (SMT) — After examination by a qualified Doctor of Chiropractic (DC), a SMT intervention consisting of up to 10 sessions over 3 months will be designed focusing on spinal manipulation and/or mobilization of the lower thoracic, lumbar and/or sacroiliac joints. Adjunctive use of myofascial and/or stretching techniques are allowed as they are commonly used along with SMT, and can be considered a standard accompaniment to SMT.
  Arms: Spinal Manipulation Therapy (SMT)
Procedure: Yoga — The Yoga for Veterans with cLBP program consists of up to 10 weekly, 60-minute instructor-led sessions along with 15-20 minutes of yoga practiced at home each non-session day. The initial session is 75 minutes (15 minutes longer than the other sessions). The yoga program can be considered classical hatha yoga with influences from Iyengar and Viniyoga yoga. These styles emphasize modifications and adaptations including the use of props such as straps and blocks to minimize the risk of injury and make the poses accessible to people with health problems and limitations (Iyengar, 1979). The instructor leads participants through a series of 23 yoga poses (32 total variations) at a slow-moderate pace.
  Arms: Yoga

SUMMARY:
VETERANS ONLY. Chronic low back pain (cLBP) is common. Most Americans will have at least one episode of low back pain in their lifetimes. Approximately 50% of all US Veterans have chronic pain, and CLBP is the most common type of pain in this population. This study will use a sequential randomized, pragmatic, 2-step comparative effectiveness study design. The main goal is to identify the best approach for treating cLBP using commonly recommended non-surgical and non-pharmacological options. The first step compares continued care and active monitoring (CCAM) to internet-based pain self-management (Pain EASE) and an enhanced physical therapy intervention that combines Pain EASE with tailored exercise and physical activity. Patients who do not have a significant decrease in pain interference (a functional outcome) in Step 1 and those desiring additional treatment will be randomized in Step 2 to yoga, spinal manipulation therapy (SMT), or therapist-delivered cognitive behavioral therapy (CBT). Participants proceeding to randomization in Step 2 will be allowed to exclude up to one of the three Step 2 treatments based on their preferences. The investigators' primary hypothesis for the first treatment step is that an enhanced physical therapy intervention that combines pain self-management education with a tailored exercise program will reduce pain interference greater than internet-based pain self-management alone or CCAM in Veterans with cLBP. The primary outcome is change in pain interference at 3 months, measured using the Brief Pain Inventory (BPI) pain interference subscale. Study participants will be followed for one year after initiation of their final study treatments to assess the durability of treatment effects. The study plans to randomize 2529 patients across 20 centers.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is common. The point prevalence of low back pain in the US is about 25%, and the majority of Americans will have at least one episode of low back pain in their lifetimes. Approximately 50% of all US Veterans have chronic pain, and cLBP is the most common type of pain in this population. Low back pain is the second most common condition leading patients to seek a physician's care. In addition, cLBP is costly. Healthcare expenditure for low back pain in the US is greater than $30 billion per year, and total expenditures including the cost of disability approach $100 billion per year. In fact, low back pain is the most common cause of work-related disability and is a major cause of service- connected disability amongst US Veterans. Making matters worse, the US is in the midst of a growing opioid abuse epidemic having its roots in the lack of understanding of how to effectively treat cLBP and other common forms of acute and chronic pain.

Using a sequential randomized, pragmatic, 2-step comparative effectiveness study design, the main goal is to identify the optimal approach to cLBP treatment employing commonly recommended non-surgical, non-pharmacological options. Options for treatment in this trial were selected based on the VA's stepped-care model for the treatment of chronic pain, availability of treatments, controversies in current clinical practice, and the surveyed preferences of both Veterans with cLBP and VA healthcare providers. The implementation of study results has been kept closely in mind, and stakeholder input has been incorporated.

The first step compares continued care and active monitoring arm (CCAM) to internet-based pain self-management (Pain EASE) and an enhanced physical therapy intervention that combines Pain EASE with tailored exercise and physical activity. The utility of tailored exercise requiring physical therapist guidance added to internet-based self-management has not been examined. A CCAM arm is included in this step to definitively assess the effectiveness of these initial treatment options. Patients failing to achieve clinically significant reductions in pain interference (a functional outcome) in Step 1 and those desiring additional treatment will be randomized in Step 2 to yoga, spinal manipulation therapy (SMT), or therapist-delivered cognitive behavioral therapy (CBT). These options appear in consensus guidelines although little information is available to help patients and providers select the most effective option. Each option has a distinct theoretical basis for effectiveness with yoga described as a mind-body therapy, SMT as a technique to adjust the structural relationships of the spine, and CBT as a psychological or behavioral approach. While the literature suggests approximate clinical equipoise between these treatments, costs, side effects, access to specific options and patient/provider acceptance may differ significantly. Participants proceeding to randomization in Step 2 will be allowed to exclude up to one of the three Step 2 treatments based on their preferences.

The investigators' primary hypothesis corresponding to the first treatment step is that an enhanced physical therapy intervention that combines pain self-management education with a tailored exercise program will reduce pain interference greater than internet-based pain self-management alone or CCAM in Veterans with cLBP. For the second step, the study has been powered to detect clinically meaningful pairwise differences among the three treatments. The primary outcome is change in pain interference at 3 months, measured using the Brief Pain Inventory (BPI) pain interference subscale. This is a widely accepted functional outcome in musculoskeletal pain trials and emphasizes an endpoint important to patients, providers and healthcare management systems. Study participants will be followed for one year after initiation of their final study treatments to assess the durability of treatment effects.

The investigators will leverage the power of this large study and maximize its impact by incorporating additional outcome measures as recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consortium and other pain trials consensus groups. These secondary outcomes include pain severity, physical functioning, depression, anxiety, fatigue, sleep, global impression of change, and quality of life. The investigators will evaluate the impact of patient characteristics, treatment preferences and expectations on study outcomes as these variables have been identified in smaller studies to modify treatment response. To derive information rapidly translatable to changes in VA care, the investigators will collect information critical for implementation of the treatment strategies under study. Key implementation factors will include treatment fidelity, treatment adherence, patient acceptance, provider acceptance, logistical feasibility, and resource requirements. Finally, a carefully designed costs and downstream budget impact aim will provide additional practical information for clinical managers and policy makers related to non-pharmacological treatments for cLBP.

The study will involve diverse VA centers with respect to geographical region, racial characteristics of the population served and facility size. The study plans to randomize 2529 patients across 20 centers. Preliminary site surveys indicate a high level of enthusiasm for the project. In addition, a query of the VA's Corporate Data Warehouse (CDW) identified more than 850,000 potential cLBP study subjects receiving regular care through VA. Twenty-five VA medical centers have more than 10,000 potentially eligible patients underscoring the high prevalence of cLBP. The investigators' pragmatic trial design will incorporate broad eligibility criteria.

Chronic low back pain is an enormous problem for the VA, the United States and many other countries. This study will provide definitive information concerning the effectiveness, costs, acceptability, and implementation of several commonly used, patient-preferred, non-pharmacological treatment options. All the selected treatment options carry relatively low levels of risk, are guideline congruent, and are consistent with stepped-care models of healthcare delivery used by the VA and other healthcare organizations. The impact on VA healthcare is expected to be large and immediate.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Low back pain

   1. present for at least 6 months,
   2. present most days or everyday,
   3. interferes the most with activities considering all of the places where the patient experiences pain;
2. Pain, Enjoyment, General Activity (PEG) score of 4 or greater;
3. Veteran age 18 years or older, either sex, any racial or ethnic background;
4. Able to comprehend and willing to sign the study informed consent form;
5. Able to attend in-person treatment sessions;
6. Anticipate continuing care at the enrolling VA for the period of the study;
7. Stable access to the internet at home, work, or other location (e.g. mobile phone), and an email address.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Currently enrolled in any other interventional study unless exempted by CSP;
2. Acute or chronic illness that would prevent the Veteran from receiving study treatments offered (e.g., uncontrolled hypertension, recent myocardial infarction within the last 6 months, unstable angina, acute congestive heart failure);
3. Neurological impairment related to disease of the spine or other causes preventing participation in any of the treatment modalities under study;
4. Current or recent (last 3 months) treatment involving Cognitive Behavioral Therapy, Spinal manipulation therapy, or Yoga;
5. Current severe alcohol or substance abuse use disorder;
6. Severe psychiatric illness (e.g. current psychosis, current suicidal ideation, or psychiatric illness requiring hospitalization within the last 6 months);
7. Undergoing evaluation for back surgery or planned back surgery;
8. Cognitive or severe hearing or visual impairment preventing participation in treatment options or outcome measure assessments;
9. Pregnancy;
10. Refusal to provide written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2529 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Interference scale | 3 months post-treatment
  Pain interference will be assessed with the Brief Pain Inventory (BPI) Interference subscale, a validated measure that rates pain interference of pain on 7 items (mood, physical activity, work, social activity, relations, sleep, and life enjoyment). BPI scores range 0 to 10, with higher scores representing worse pain interference, and a 1-point change considered clinically important. Linear mixed effects models will be used to compare the primary outcome (change in pain interference score from pre-treatment to 3 months after treatment) between Step 1 treatments in all participants and between Step 2 treatments in Step 1 non-responders. The mixed effects model will include treatment and study site as fixed effects, and therapist as random effects. For the comparison of Step 1 treatments, the model will also include a fixed effect for opioid use at study entry.

SECONDARY OUTCOMES:
Serious Adverse Events | 3, 6, 9, and 12 months post-treatment
  Attributable and possibly attributable serious adverse events
Brief Pain Inventory (BPI) Interference scale | 6, 9, and 12 months post-treatment
  Pain interference will be assessed with the Brief Pain Inventory (BPI) Interference subscale, a validated measure that rates pain interference of pain on 7 items (mood, physical activity, work, social activity, relations, sleep, and life enjoyment). BPI scores range 0 to 10, with higher scores representing worse pain interference, and a 1-point change considered clinically important.
Patient Health Questionnaire-9 (PHQ-9) | 3, 6, 9, and 12 months post-treatment
  This is a tool to measure comorbid depression. This scale is frequently used in VA settings, has been well validated, and is a quick self-administered questionnaire.
  - Possible range for PHQ-9 is 0-27. Higher scores indicate more severe depression. 0-4: None/Minimal depression, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, 20-27: Severe depression.
Numeric Rating Scale (NRS) | 3, 6, 9, and 12 months post-treatment
  Possible range of NRS is 0 to 10 with higher scores reflecting greater perceived pain.
Roland-Morris Disability Questionnaire (RMDQ) | 3, 6, 9, and 12 months post-treatment
  Roland-Morris Disability Questionnaire (RMDQ) measures low-back specific physical function. The RMDQ consists of 24 statements (e.g., "I stay at home most of the time because of my back and/or leg pain") that respondents simply endorse "yes" or "no."
  - Possible range of RMDQ is 0-24 with higher scores reflecting greater perceived disability.
Generalized Anxiety Disorder-7 Scale (GAD-7) | 3,6, 9, and 12 months post-treatment
  This is a self-administered tool to assess anxiety.
  - Possible range for GAD-7 is 0-21. Higher scores indicate more severe anxiety symptoms. 0-4: None/Minimal anxiety; 5-9: Mild Anxiety; 10-14: Moderate Anxiety; 15-21: Severe anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep | 3, 6, 9, and 12 months post-treatment
  Patient-Reported Outcomes Measurement Information System (PROMIS) 4-item sleep scale assesses perceptions of sleep quality, sleep depth, and restorative sleep.
  - Possible range for PROMIS 4-item sleep scale is 4 to 20. The scale has five response options (e.g., 1 = not at all to 5 = very much) with higher scores indicating more sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue | 3, 6, 9, and 12 months post-treatment
  To assess fatigue, the PROMIS 4-item fatigue scale will be used. Possible range for PROMIS 4-item fatigue scale is 4-20. The scale has five response options (e.g., 1 = not at all to 5 = very much), with higher scores indicating worse fatigue.
Global Mental Health (GMH-2) | 3, 6, 9, and 12 months post-treatment
  To assess mental health, the two-item Global Mental Health (GMH-2) scale will be used. Possible range for GMH-2 is 2-10. The scale has five response options (e.g. 1 = excellent to 5 = poor), with higher scores indicating worse mental health.
Global Physical Health (GPH-2) | 3, 6, 9, and 12 months post-treatment
  To assess physical health, the two-item Global Physical Health (GPH-2) scale will be used. Possible range for GPH-2 is 2-10. The scale has five response options (e.g. 1 = excellent to 5 = poor), with higher scores indicating worse physical health.
Patient Global Impression of Change (PGIC) | 3,6, 9, and 12 months post-treatment
  This is a single-item 7-point scale that captures a patient's rating of overall improvement.
EuroQol Quality of Life Scale (EQ-5D-5L) | 3, 6, 9, and 12 months post-treatment
  This is a 5-question generic health status measure to assess level of impairment in mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In addition, the scale has a 20cm Visual Analog Scale to assess overall self-rated health status.
Non-VA Healthcare Utilization | 3, 6, 9, and 12 months post-treatment
  medical care obtained outside of the VA
Societal Cost | 3, 6, 9, and 12 months post-treatment
  overall costs to the participant and others
Follow-up Treatments and Medications | 3, 6, 9, and 12 months post-treatment
  medications and non-study treatment for back pain

CONTACTS AND LOCATIONS:
Overall Officials: David J Clark, PhD MD, Study Chair — VA Palo Alto Health Care System, Palo Alto, CA; Matthew J. Bair, MD MS, Study Chair — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (19):
- United States (19):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, North Las Vegas, Nevada
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark JD, Bair MJ, Belitskaya-Levy I, Fitzsimmons C, Zehm LM, Dougherty PE, Giannitrapani KF, Groessl EJ, Higgins DM, Murphy JL, Riddle DL, Huang GD, Shih MC. Sequential and Comparative Evaluation of Pain Treatment Effectiveness Response (SCEPTER), a pragmatic trial for conservative chronic low back pain treatment. Contemp Clin Trials. 2023 Feb;125:107041. doi: 10.1016/j.cct.2022.107041. Epub 2022 Dec 7. PMID 36496154